CLINICAL TRIAL: NCT03949530
Title: IDL-2965 - A Phase I, Randomized, Double-blind, Placebo-controlled, Single and Multiple Oral Dose, Safety, Tolerability, and Pharmacokinetic Study in Healthy Subjects and Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Study of Safety & Blood Levels of IDL-2965 in Healthy Subjects and Patients With a Special Type of Pulmonary Fibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to development challenges associated with the SARS-CoV-2 pandemic and emerging nonclinical data
Sponsor: Indalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: Indalo (IDL)-2965-IPF-001; 2019-000173-23 (EudraCT Number)
Record Dates: First submitted 2019-05-06; First posted 2019-05-14 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IDL-2965 Oral Capsule (Experimental): IDL-2965 oral capsule, single and multiple doses
  Interventions: Drug: IDL-2965 Oral Capsule
- Placebo Oral Capsule (Placebo Comparator): Placebo oral capsule, single and multiple doses
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: IDL-2965 Oral Capsule — Investigational drug
  Arms: IDL-2965 Oral Capsule
Drug: Placebos — Placebo
  Arms: Placebo Oral Capsule

SUMMARY:
The purpose of this study is to test the safety and tolerability of the drug candidate IDL-2965 and to see how it is absorbed, processed, and removed by the body.

DETAILED DESCRIPTION:
IDL-2965 is an oral integrin antagonist antifibrotic being studied as a potential treatment for IPF and Nonalcoholic Steatohepatitis (NASH). This double-blind, randomized, placebo-controlled, single and multiple oral dose study will be conducted in 3 parts. Part A will comprise a single-dose, sequential-group design in healthy subjects, incorporating a food-effect evaluation. Part B will consist of a multiple-dose, sequential-group design in healthy subjects. Part C will be a multiple-dose, sequential-group design in subjects with IPF.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

• Male and female subjects aged between 18 and 60 years, with a body mass index between 18.0 and 32.0 kg/m2.

IPF subjects:

* Male and female subjects over 40 years of age.
* Diagnosis of idiopathic pulmonary fibrosis
* Idiopathic pulmonary fibrosis has been stable for at least 3 months.

Exclusion Criteria:

Healthy subjects and IPF subjects:

* Significant history or clinical manifestation of any disease/disorder, other than IPF.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound
* Poor peripheral venous access
* Use or intend to use any medications, tobacco or nicotine containing products or electronic cigarettes.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs

IPF subjects:

• Pulmonary function tests and other diagnostic procedures inconsistent with diagnosis of idiopathic pulmonary fibrosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent Adverse Events (AEs), AEs leading to discontinuation from Investigational Medicinal Product (IMP) or the study, serious adverse events (SAEs), and deaths. | Single Ascending Dose (SAD): up to 7 Days/ Multiple Ascending Dose (MAD): up to 21 Days/ IPF MAD: up to 40 Days
  Safety

SECONDARY OUTCOMES:
Pharmacokinetic (PK) | SAD: up to 7 Days / MAD: up to 21 Days / IPF MAD: up to 40 Days
  Area under the plasma concentration-time curve from time zero to 24 hours

OTHER OUTCOMES:
Exploratory Pharmacodynamic (PD) | SAD: up to 7 Days / MAD: up to 21 Days / IPF MAD: up to 28 Days
  Change from baseline in phosphorylated small mothers against decapentaplegic (pSMAD) from bronchoalveolar lavage fluid cells

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MRCS FFPM, Study Director — Indalo Therapeutics, Inc.
Locations (1):
- Covance CRU, Leeds, United Kingdom